CLINICAL TRIAL: NCT07202429
Title: Additive Role of Mean Apparent Diffusion Coefficient (ADCmean) Value Measurements to the Ovarian-Adnexal Reporting and Data System (O-RADS) MRI Score in Stratifications of Adnexal Lesions
Brief Title: Additive Role of ADC Value to ORADS in Adnexal Lesions
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Badawy, Lecturer of Radiology, Cairo University, Cairo University
Other Study IDs: mri dwi in adnexal lesions
Record Dates: First submitted 2023-09-06; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Neoplasms
Keywords: MRI-ORADS; ADC value; Ovarian neoplasms
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Benign Adnexal Lesions: Description: Participants with adnexal lesions that were confirmed as benign on histopathology.
  Description: Dynamic MRI imaging including diffusion-weighted imaging (DWI) and apparent diffusion coefficient (ADC) measurement, used for lesion characterization with O-RADS scoring.
  Interventions: Device: MRI
- Borderline adnexal lesions: Description: Participants with adnexal lesions that were confirmed as borderline on histopathology.
  Description: Dynamic MRI imaging including diffusion-weighted imaging (DWI) and ADC measurement, used for lesion characterization with O-RADS scoring.
  Interventions: Device: MRI
- Malignant adnexal lesions: Description: Participants with adnexal lesions that were confirmed as maligannt on histopathology.
  Description: Dynamic MRI imaging including diffusion-weighted imaging (DWI) and ADC measurement, used for lesion characterization with O-RADS scoring.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — "Multiparametric MRI of adnexal lesions, including conventional sequences, diffusion-weighted imaging (DWI) with apparent diffusion coefficient (ADC) measurement, and dynamic contrast-enhanced (DCE) MRI. Imaging findings were evaluated using the O-RADS MRI scoring system."

SUMMARY:
Evaluation of the impact of adding mean apparent diffusion coefficient (ADC mean) measurements to the Ovarian-Adnexal Imaging Reporting and Data System MRI (O-RADS MRI) scoring for adnexal lesion characterization using a combined O-RADS MRI/ADC mean reading approach.

DETAILED DESCRIPTION:
The patients will be referred from the Gynecology department to the Kasr Al-Ainy Radiology department (Women's imaging unit) based on preliminary ultrasound examination used for cases selection.

Female patients with adnexal lesions on ultrasound were subjected to MRI examination, Standardised MRI sequences will used, including DWI and DCE sequences. blinded to histopathological data, according to the O-RADS MRI scoring system. A quantitative analysis method will applied by placing a ROI on the ADC maps obtained from single-exponential DWI sequences.

Additive role of ADC value will be comparied to O-RADs according to gold standard (pathological examination of adnexal lesions) after excision to correlate results of imaging and pathology.

MRI examination: MR imaging was performed using a 1.5-T magnet using torso coil Diffusion WI: with b values 0, 500, 1000 and 1500 as well as ADC map. Dynamic contrast enhanced study: using 10cc of Gadopentetate dimeglumine and 20ml of saline. Injection is manual. Examination time is 4minutes with 8 series. Scan time for each series: 32secs

ELIGIBILITY:
Inclusion Criteria:

* (1) Female patient any age with at least one adnexal lesion detected by U/S reported as O-RADS3to5.

  (2) The interval between operation and ultrasonography did not exceed 120 days. (3) Subsequent surgery with histological examination or stability at follow-up imaging for at least 1 year.

  (4) For bilateral adnexal masses, the mass with the most complex features was included.

  (5)If two masses had similar morphologies, the largest mass was included.

Exclusion Criteria:

1. Female patient any age with adnexal lesions detected by U/S reported as O-RADS1and2.
2. Cysts that were deemed to be clearly physiological and less than 3 cm in maximum diameter.
3. No histopathological findings or follow-up < one year .
4. Previous bilateral adnexectomy.
5. Contraindications to MRI examination including

   * Absolute contraindications: such as The cardiac implantable electronic device (CIED), Metallic intraocular foreign bodies, ….)
   * Relative contraindications: such as Coronary and peripheral artery stents, Ocular prosthesis,……)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: female patients any age with ovarian lesions
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Mean ADC value of adnexal lesions | March 2023 to june 2024
  Measurement of mean apparent diffusion coefficient (ADCmean) values in adnexal lesions using diffusion-weighted imaging (DWI). Unit of Measure: ADC value (×10-³ mm²/s)
Diagnostic performance of O-RADS MRI + ADC system | March 2023 to june 2024
  Evaluation of diagnostic performance (sensitivity, specificity, accuracy) of O-RADS MRI scoring combined with ADC values, compared with O-RADS MRI system alone. Unit of Measure: Percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Lamia Salah Eldin, M.D, Principal Investigator — kasr-alainy cairo university; Manar Alaa Eldin Osman, M.D, Study Director — kasr-alainy cairo university; Mohammed Aly Shalaby, M.D, Study Chair — kasr-alainy cairo university
Locations (1):
- Kasr Al-Ainy Faculty of Medicine, Cairo University, Cairo, Cairo Governorate, Egypt